CLINICAL TRIAL: NCT05354934
Title: Study of Entry and Continuation in Care for People Living With HIV in French Guiana
Acronym: EMVIH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: EMVIH
Record Dates: First submitted 2022-04-05; First posted 2022-05-02 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Human Immunodeficiency Virus
Keywords: Human Immunodeficiency Virus; french guiana; maintain in care; HIV diagnosis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People living with HIV: The questionnaire includes the following modules
  * Demography and socio-economic conditions
  * Screening and modalities of discovery and announcement of HIV infection
  * Time and modalities of introduction of antiretroviral drugs after diagnosis
  * Knowledge of HIV infection
  * The perception of follow-up in the health care service
  * Experiences of stigma
  * Barriers to accessing care
  * Periods of loss of sight and reasons for this
  * Perceived health status, mental health (PHQ4), chronic illness, functional limitations
  * Addictions
  * Social network and support
  * Clinical data Date of HIV diagnosis Date of introduction of antiretrovirals CD4 count at diagnosis Viral load at diagnosis Period without follow-up for more than 12 months CD4 nadir Last CD4 count Last viral load Antiretroviral treatment at last consultation Comorbidities Initial hospitalisation Recent hospitalization
  Interventions: Other: quetionnaire

INTERVENTIONS:
Other: quetionnaire — The questionnaire includes the following modules
  * Demography and socio-economic conditions
  * Screening and modalities of discovery and announcement of HIV infection
  * Time and modalities of introduction of antiretroviral drugs after diagnosis
  * Knowledge of HIV infection
  * The perception of follow-up in the health care service
  * Experiences of stigma
  * Barriers to accessing care
  * Periods of loss of sight and reasons for this
  * Perceived health status, mental health (PHQ4), chronic illness, functional limitations
  * Addictions
  * Social network and support
  * Clinical data Date of HIV diagnosis Date of introduction of antiretrovirals CD4 count at diagnosis Viral load at diagnosis Period without follow-up for more than 12 months CD4 nadir Last CD4 count Last viral load Antiretroviral treatment at last consultation Comorbidities Initial hospitalisation Recent hospitalization

SUMMARY:
Research Involving the Non-Interventional Human Subject (RIPH category 3). Non-interventional, cross-sectional, multicentre, descriptive and analytical epidemiological study.

A cross-sectional, pseudo-anonymous questionnaire focusing on entry and retention in care will be administered to a sample of PLHIV presenting for consultation in one of the GHT hospitals over a 12-month period.

A sample of 300 PHAs is envisaged to have sufficient power to highlight the main factors associated with periods of loss of sight.

Main objective:

- To identify factors associated with loss of sight for more than 12 months among people living with HIV in Guyana

Secondary objectives:

* To identify factors associated with a delay in the introduction of ARVs among PLHIV in Guyana
* To describe the perception of the quality of the announcement of the diagnosis of HIV
* To describe the difficulties encountered by PLHIV during their hospital follow-up in French Guyana
* To assess the perceived stigma associated with HIV and its consequences in daily life

DETAILED DESCRIPTION:
French Guyana is the French territory most affected by the HIV epidemic, with a prevalence estimated at between 1.13 and 1.18% of the adult population aged 15 to 49, and the incidence remains high at 0.90 per 1,000 people in 2018(1,2). Although French Guyana is a territory where the rate of screening per inhabitant is high, the proportion of infections diagnosed at a very advanced stage remains stable (from 30% in Cayenne to 45% in Saint-Laurent-du-Maroni). HIV/AIDS remains one of the main causes of premature mortality in French Guyana, with serious opportunistic pathologies specific to the territory, such as disseminated histoplasmosis.

The context of the discovery of HIV infection, the quality of the ensuing announcement and the time taken to introduce antiretroviral treatment are important determinants of the care pathway and the subsequent management in the "test and treat" era. Regular medical follow-up, good understanding of one's infection and good adherence to treatment allow the achievement of an undetectable viral load, immune restoration, maintenance of good health and reduction of the risk of secondary transmission (3, 4, 5)(3-5).

In 2018, the cascade of care in Guyana was estimated at 90% of PLHIV diagnosed, 91% of patients screened on treatment, and 94% of patients on antiretroviral treatment for more than 6 months in treatment success(1).

The WHO sets "Test and Treat" targets at 7 days following serological diagnosis in the absence of medical contraindication(6), or even the same day in circumstances where access to consultations is difficult. However, the median time for introducing antiretrovirals (ARVs) in French Guyana was estimated at 22 days in 2019(7), far from the 7-day target. This average delay, which is key to controlling the epidemic, has not been the subject of further analysis of its determinants. Territorial disparities are already apparent, with a longer delay in the west than on Cayenne Island (24 days at the West Guyana Hospital Centre and 20 days at the Cayenne Hospital Centre)(7).

On the other hand, the rate of LOS is high in French Guyana and particularly in Saint Laurent du Maroni where it is estimated that between 2 and 11% of people are lost to follow-up each year (1).

In this context, delays in the introduction of antiretroviral treatment and the risk of loss of sight (LOS) among PLHIV are major issues in the fight against the epidemic, both in terms of preventing progression to the AIDS stage, which is still all too common in French Guyana, and in preventing secondary transmission.

Thus, a better understanding of the quality of the diagnostic announcement will enable work to be carried out on the points that need to be improved in order to ensure effective retention in care. In the same way, by identifying the obstacles to the rapid implementation of ARVs, study team will work to remove these obstacles and provide the necessary responses to reduce the delay.

The investigators hypothesise that the increase in the rate of people lost to follow-up over time in French Guyana is associated with an increase in the social difficulties encountered by PLHIV in a context of demographic and migratory progression and a tension between the players, the fragility of the specialised care offer over time, and a possible increase in follow-up in the city, which escapes the hospital surveillance data.

Main objective:

- To identify factors associated with loss of sight for more than 12 months among people living with HIV in Guyana

Secondary objectives:

* To identify factors associated with a delay in the introduction of ARVs among PLHIV in Guyana
* To describe the perception of the quality of the announcement of the diagnosis of HIV
* To describe the difficulties encountered by PLHIV during their hospital follow-up in French Guyana
* To assess the perceived stigma associated with HIV and its consequences in daily life

Research Involving the Non-Interventional Human Subject (RIPH category 3). Non-interventional, cross-sectional, multicentre, descriptive and analytical epidemiological study.

A cross-sectional, pseudo-anonymous questionnaire focusing on entry and retention in care will be administered to a sample of PLHIV presenting for consultation in one of the GHT hospitals over a 12-month period.

A sample of 300 PHAs is envisaged to have sufficient power to highlight the main factors associated with periods of loss of sight.

The identification of factors associated with a delay in starting antiretrovirals, periods of loss of sight, as well as obstacles and facilitators to retention in care will enable local actors to recognise patients requiring particular support for continuity of care and the COREVIH's loss of sight working group, which is being set up at the same time, to work on adapted responses that are co-constructed with all the actors. It will also allow for the adaptation and development of follow-up strategies, for example through better collaboration between the hospital and the town, or with border countries.

A better understanding of the period between serological diagnosis and the initiation of ARVs among PLHIV in French Guyana will enable the tools for controlling the epidemic to be adapted, bringing us closer to the WHO's objectives, and will help to reduce the morbidity and mortality of patients through individual care adapted to the various reference centres in French Guyana.

ELIGIBILITY:
Inclusion Criteria:

* People living with HIV
* Aged 18 years and over
* Followed in one of the 3 GHT Guiana hospitals (Cayenne, Kourou, Saint-Laurent-du-Maroni)
* Not opposed to participating in the study

Exclusion Criteria:

* Be under 18 years of age
* Not be living with HIV
* Not being followed in one of the GHT Guyana hospitals
* Have a physical or mental disability that prevents them from answering the questionnaire
* Be under guardianship or under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cross-sectional, pseudo-anonymous questionnaire, focusing on entry and retention in care, will be administered to a sample of PLHIV presenting for consultation in the three GHT hospitals.
  The questionnaire will be offered once to each eligible PLHIV consulting one of the three study hospitals and not opposed to participation over a 12-month period. Inclusion will be carried out by the consulting physician or intern who will be responsible for presenting the study, collecting non-opposition and administering the questionnaire presented in paper format. The questionnaire may be completed by the qualified persons listed on the study task sheet.
  The questionnaire will be administered to a sample of the active file based on the availability of qualified persons (doctors and interns) participating in the survey. Depending on the number of subjects required, it is expected that 300 questionnaires can be administered over the study period.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-03-23 (Estimated); Study Completion 2024-06-23 (Estimated)

PRIMARY OUTCOMES:
Identifying factors associated with loss of sight for more than 12 months among people living with HIV in Guyana | more than last 12 months
  Socio-demographic, clinical, biological and therapeutic factors associated with a period of loss of sight of PLWH in Guyana. Loss of sight is defined as a period of 12 months or more of follow-up since the last specialist hospital consultation in one of the three participating hospitals.

SECONDARY OUTCOMES:
Identifying factors associated with a delay in the introduction of ARVs among PLHIV in French Guyana | baseline
  Socio-demographic, clinical, biological and therapeutic factors associated with a delay in the introduction of antiretroviral treatment for PLHIV in French Guyana. Delayed initiation of antiretroviral treatment is defined as initiation of antiretroviral drugs more than 30 days after the discovery of HIV infection when it occurred in France or Guyana and after 2013
Describe the perceived quality of the HIV diagnostic announcement with a specific questionnaire | baseline
  perceived quality of the HIV diagnostic announcement with a specific questionnaire
describe the difficulties encountered by PLHIV during their hospital follow-up in French Guyana with a specific questionnaire | baseline
  difficulties encountered by PLHIV during their hospital follow-up in French Guyana with a specific questionnaire
Assessing perceived HIV-related stigma and its impact on daily life with a specific questionnaire | baseline
  perceived HIV-related stigma and its impact on daily life with a specific questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, France, French Guiana

IPD SHARING:
Plan to Share IPD: No